CLINICAL TRIAL: NCT04789395
Title: Clinical Determination of Patients Who Intersive Care Unit and Clinical Ttreatments Have Finished Receive Ozonetheraphy With Thorax Tomography Regarding to Interstisial Fibrosis
Brief Title: Evaluation of Post-covid 19 Patients Who Receive Ozonetheraphy With Thorax CT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SİBEL BEKTAŞ, director, Gaziosmanpasa Research and Education Hospital
Other Study IDs: 08.092.r1.125
Record Dates: First submitted 2021-03-08; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Ozone Therapy for Covid 19 Pneumonia Patients
Keywords: ozone; COVİD 19; pulmonary fibrosis
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is known that enhances wound healing by oxidative stress and supports immune system besides it is cheap and has not any side effects. Aim of the study is to prevent pulmonary fibrosis by using ozone therapy as a supportive therapy on the patients who have pneumonia and ground glass opacity on thorax CT both in ICU and wards. Patients will follow for a year.

DETAILED DESCRIPTION:
The patients accepted with the diagnosis of pneumonia in Gaziosmanpaşa TREH, both in ICU and wards have treated with additional ozone therapy beside the normal treathments. In these patients the findings like ground glass opacity in thorax CT regarding to covid 19 were progressed or non changed. In the concern of these opacities turn to pulmonary fibrosis, ozone therapy has used to prevent this undesirable effect. It is known that enhances wound healing by oxidative stress and supports immune system besides it is cheap and has not any side effects.

25 patients included this study. The patients were diagnosed with Covid-19 pneumonia and treated with ozone therapy in intensive care unit and ward. After treatment was done, findings of at least %20-25 ground-glass opacity on thorax ct were the main criteria for enrollment.

The patients' follow-up program time after hospital discharge will be on 1st, 3rd, 6th and 12th month. They will continue to recieve ozon therapy once in a month during one year follow up. Ground-glass opacity rate of thorax ct scan will be recorded as less then %25, %25-50, %50-75 and above %75. Tomographies will be compared with each other and also last thorax ct before hospital discharge. These tomographies will be applied under 80 KV and this will give %40 less dosage according to routine 120 KV scans. If there is an increase in ground-glass opacities compared to the previous one, the scan will be done again on prone position and suspected lesions will be reevaluated. The pulmonary fibrosis findings of the scan will be diagnosed by a well trained radiology doctor. The evaluation of dyspnea will also done during follow-ups. mMRC(medical research council) dyspnea scale will be used for dyspnea status. SpO2 values in room-air will also recorded. FEV1, FVC and FEV1/FVC values will also be recorded to demonstrate respiratory functions.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years covid 19 pneumonia patients who have ground glass opacity on thorax CT, receiving ozone as adjuvant therapy.

Exclusion Criteria:

* pregnant patients patients who doesnt treated with ozone(hyperthyroid,pulmonary hypertension, right ventricule failure,glucose 6 P dehydrogenase defficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 patients over 18 years of age, treated with ozone in ICU and wards
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
prevention of pulmonary fibrosis in covid 19 pneumonia patients with ozone therapy | 1 year
  Ozone as an additional therapy can reduce the fibrosis

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa TREH, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)